CLINICAL TRIAL: NCT01772368
Title: A Six-Period Crossover, Dose-Ranging Study to Evaluate the Efficacy and Safety of Four Doses of FS Spiromax (Fluticasone Propionate/Salmeterol Xinafoate Inhalation Powder) Administered as Single Doses Compared With Single Doses of Fluticasone Propionate Spiromax and Open Label Advair Diskus in Adult and Adolescent Subjects With Persistent Asthma
Brief Title: Dose Ranging Study of the Salmeterol Component of Fluticasone /Salmeterol Spiromax Compared to Fluticasone Spiromax and Advair Diskus in Asthma Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FSS-AS-201
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma; dry powder inhaler; long-acting beta2-agonist; bronchodilation; bronchodilator; metered dose inhaler; inhaled corticosteroid
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination; Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- FS MDPI 100/6.25 mcg (Experimental): Subjects inhaled a single dose of 100 mcg fluticasone propionate and 6.25 mcg salmeterol xinafoate.
  Interventions: Drug: FS MDPI; Drug: Albuterol
- FS MDPI 100/12.5mcg (Experimental): Subjects inhaled a single dose of 100 mcg fluticasone propionate and 12.5 mcg salmeterol xinafoate.
  Interventions: Drug: FS MDPI; Drug: Albuterol
- FS MDPI 100/25 (Experimental): Subjects inhaled a single dose of 100 mcg fluticasone propionate and 25 mcg salmeterol xinafoate.
  Interventions: Drug: FS MDPI; Drug: Albuterol
- FS MDPI 100/50 (Experimental): Subjects inhaled a single dose of 100 mcg fluticasone propionate and 50 mcg salmeterol xinafoate.
  Interventions: Drug: FS MDPI; Drug: Albuterol
- Fp MDPI 100 mcg (Active Comparator): Subjects inhaled a single dose of 100 mcg fluticasone propionate.
  Interventions: Drug: Fp MDPI; Drug: Albuterol
- Advair Diskus 100/50 mcg (Active Comparator): Subjects inhaled a single dose of 100 mcg fluticasone propionate and 50 mcg salmeterol xinafoate. This arm is the only arm which is open-label because the inhaler device was different than the MDPI used in the other treatment arms.
  Interventions: Drug: Advair Diskus; Drug: Albuterol

INTERVENTIONS:
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  Fp at 100 mcg was an active comparator (single dose). Further, participants were instructed to administer two inhalations of Fp MDPI 50 mcg twice daily (100 mcg total dose) during the Run-in (to replace the participant's current inhaled corticosteroid) and Washout Periods between treatments.
  Other Names: fluticasone propionate; inhaled corticosteroid; Fp Spiromax
  Arms: Fp MDPI 100 mcg
Drug: FS MDPI — FS MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate and salmeterol xinafoate dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened. The fluticasone propionate component was a fixed dose of 100 mcg. The salmeterol xinofoate dosage varied: 6.25, 12.5, 25 or 50 mcg.
  Other Names: fluticasone propionate; inhaled corticosteroid; Salmeterol xinafoate; β2 adrenoceptor agonist; FS Spiromax
  Arms: FS MDPI 100/12.5mcg; FS MDPI 100/25; FS MDPI 100/50; FS MDPI 100/6.25 mcg
Drug: Advair Diskus — ADVAIR DISKUS (100/50 mcg fluticasone propionate/salmeterol xinafoate) consists of a dry powder formulation of fluticasone propionate and salmeterol xinafoate in a lactose excipient. The dry powder is contained within individual blisters on a double foil strip within the device. Activation of the device opens a single blister of medication which is then dispersed into the air-stream by patient inhalation.
  Other Names: fluticasone propionate; inhaled corticosteroid; salmeterol xinafoate; β2 adrenoceptor agonist
  Arms: Advair Diskus 100/50 mcg
Drug: Albuterol — Albuterol (Pro-Air) hydrofluoroalkane (HFA) metered dose inhaler (MDI), was provided to be used as needed for the relief of asthma symptoms during both the run-in and treatment periods (to replace the subject's current rescue medication).
  Other Names: Pro-Air; short-acting β2-adrenergic agonists

SUMMARY:
The primary objective of this study is to evaluate the dose response, efficacy, and safety of 4 different doses of salmeterol Spiromax (6.25, 12.5, 25, and 50 mcg) each combined with a fixed dose of fluticasone propionate (100 mcg) delivered as Fluticasone/Salmeterol Spiromax® Inhalation Powder (FS Spiromax) when administered as a single dose in subjects 12 years of age and older with persistent asthma.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind and open-label active-controlled, single-dose, 6 period crossover, dose-ranging study conducted in male and female subjects ages 12 years and older with persistent asthma.

Fluticasone propionate multidose dry powder inhaler (Fp MDPI) 50 mcg was provided (to replace the subject's current inhaled corticosteroid (ICS)) throughout the 14 day run-in period and each of the washout periods between treatments. Subjects were instructed to administer 2 inhalations of Fp MDPI 50 mcg (100 mcg total dose) twice daily during the run-in and washout periods. All other medications for the treatment of asthma were discontinued at or prior to the screening visit.

A short-acting β2-adrenergic agonist (SABA), salbuterol HFA, MDI, was provided (to replace the subject's current rescue medication) for symptomatic relief of asthma symptoms in each the run-in, treatment, and washout periods.

Treatment period lasted 5 weeks with a 5 to 7 day washout between each of the six single dose treatments:

* fluticasone propionate/salmeterol xinafoate multidose dry powder inhaler (FS MDPI) given in doses of 6.25, 12.5, 25, or 50 mcg of salmeterol xinafoate in blinded fashion.
* fluticasone propionate multidose dry powder inhaler (Fp MDPI) 100 mcg in blinded fashion
* ADVAIR DISKUS, 100/50 mcg in open-label fashion

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* General good health
* Diagnosis of asthma as defined by the National Institutes of Health (NIH)
* A best FEV1 of 40%-85% of the predicted normal value during the screening visit (SV)
* Subjects need to demonstrate a ≥ 15% reversibility of FEV1 within 30 minutes following 4 inhalations of albuterol inhalation aerosol (if required, spacers are permitted for reversibility testing) at the SV.
* Other inclusion criteria apply

Exclusion Criteria:

* History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks prior to the SV.
* Any asthma exacerbation requiring oral corticosteroids within 3 months of the SV. A subject must not have had any hospitalization for asthma within 6 months prior to the SV.
* Taking long-acting β-agonists within 2 weeks of the SV
* Other exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Teva Investigational Site 10453, Denver, Colorado
  - Teva Investigational Site 10452, North Dartmouth, Massachusetts
  - Teva Investigational Site 10455, St Louis, Missouri
  - Teva Investigational Site 10454, Skillman, New Jersey
  - Teva Investigational Site 10448, Raleigh, North Carolina
  - Teva Investigational Site 10451, Medford, Oregon
  - Teva Investigational Site 10449, Portland, Oregon
  - Teva Investigational Site 10457, El Paso, Texas
  - Teva Investigational Site 10450, New Braunfels, Texas
  - Teva Investigational Site 10456, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 105 subjects with asthma were screened for this study. Of the 105 subjects screened, 82 subjects at 10 investigational sites in the US met entry criteria and were considered to be eligible to enter the run-in period.
Pre-assignment Details: Ten subjects failed randomization.
Groups:
- All Participants: All subjects, regardless of the order of treatments to which they were randomized in this cross-over study.
Period: Overall Study
Arm/Group | All Participants
Started | 72
Received Fp MDPI 100 mcg | 67
Received FS MDPI 100/6.25 mcg | 68
Received FS MDPI 100/12.5mcg | 69
Received FS MDPI 100/25 mcg | 67
Received FS MDPI 100/50 mcg | 68
Received Advair Diskus 100/50 mcg | 66
Completed | 65
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population
Arm/Group | All Participants
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64
  Black | 7
  Other | 1
Weight [Mean (Standard Deviation); unit: kg] | 79.2 (14.17)
Height [Mean (Standard Deviation); unit: cm] | 170.0 (9.76)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (3.35)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-Adjusted Area Under the Curve For Forced Expiratory Volume In 1 Second Over 12 Hours Post-dose (FEV1 AUC0-12)
Description: Standardized baseline-adjusted FEV1 AUC0-12 was defined as the area under the curve for baseline-adjusted FEV1 measurements from the predose to 12 hours postdose time points using the trapezoidal rule based on actual (not scheduled) time of measurement and was standardized by dividing the actual time of last non-missing FEV1 measurement. Baseline-adjusted FEV1 was calculated as postdose FEV1 after subtracting period-specific baseline FEV1. The period-specific baseline FEV1 was measured at predose within 5 minutes of AM dose administration at each treatment visit. If that value was missing, then FEV1 measured at 30 minutes predose was used as the period-specific baseline.
Time Frame: Pre-dose: 30 minutes prior, within 5 minutes of dose. Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 9, 12 hours
Population: The full analysis set (FAS) included all subjects in the ITT population who received at least 1 dose of study drug and had at least 1 evaluable standardized baseline-adjusted FEV1 AUC0-12.
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- FS MDPI 100/25 mcg: Subjects inhaled a single dose of 100 mcg fluticasone propionate and 25 mcg salmeterol xinafoate.
- FS MDPI 100/50 mcg: Subjects inhaled a single dose of 100 mcg fluticasone propionate and 50 mcg salmeterol xinafoate.
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg
Number analyzed (Participants) | 67 | 68 | 69 | 67 | 68 | 66
mL | 52.13 (38.071) | 203.84 (38.072) | 248.98 (38.025) | 279.69 (38.121) | 303.43 (38.062) | 245.56 (38.148)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/6.25 mcg vs FS MDPI 100/12.5mcg vs FS MDPI 100/25 mcg vs FS MDPI 100/50 mcg; A linear in log-dose-trend contrast was constructed to evaluate the dose-response trend, where the logarithm of dose was defined precisely as log (dose+1) to accommodate the case of Fp MDPI 100 mcg, since the dose used in this trend analysis was the salmeterol dose. The study was considered positive if the trend test was positive and the test involving the highest FS MDPI dose (100/50 mcg) compared with Fp MDPI 100 mcg was positive, regardless of the results of the tests for the other doses; Test type: Other — linearity statistical test; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; Fixed effects of sequence, period and treatment; a random effect of subject within sequence; and a covariate of period-specific baseline FEV1
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/50 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/50 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 251.30, 95% CI 2-sided [215.6 to 287.1] — FS MDPI 100/50 mcg - Fp MDPI 100 mcg
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/25 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/25 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 227.56, 95% CI 2-sided [191.6 to 263.5] — FS MDPI 100/25 mcg - Fp MDPI 100 mcg
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/12.5mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/512.5 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 196.85, 95% CI 2-sided [161.2 to 232.5] — FS MDPI 100/12.5 mcg - Fp MDPI 100 mcg
Statistical Analysis 5: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/6.25 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/6.25 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 151.71, 95% CI 2-sided [115.9 to 187.5] — FS MDPI 100/6.25 mcg - Fp MDPI 100 mcg
Statistical Analysis 6: Comparison: Fp MDPI 100 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between Advair Diskus 100/50 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 193.42, 95% CI 2-sided [157.4 to 229.5] — Advair Diskus 100/50 mcg - Fp MDPI 100
Statistical Analysis 7: Comparison: FS MDPI 100/50 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/50 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.0017, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 57.88, 95% CI 2-sided [22.0 to 93.7] — FS MDPI 100/50 - Advair Diskus 100/50 mcg
Statistical Analysis 8: Comparison: FS MDPI 100/25 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/25 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.0624, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 34.14, 95% CI 2-sided [-1.8 to 70.1] — FS MDPI 100/25 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 9: Comparison: FS MDPI 100/12.5mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/12.5 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.8503, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = 3.42, 95% CI 2-sided [-32.3 to 39.1] — FS MDPI 100/12.5mcg - Advair Diskus 100/50 mcg
Statistical Analysis 10: Comparison: FS MDPI 100/6.25 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between FS MDPI 100/6.25 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.0229, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = -41.72, 95% CI 2-sided [-77.6 to -5.8] — FS MDPI 100/6.25 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 11: Comparison: Fp MDPI 100 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between Fp MDPI 100 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 2 sided 0.05 level; [statistical method as in outcome 1, analysis 1]; LSM difference = -193.42, 95% CI 2-sided [-229.5 to -157.4] — Fp MDPI 100 mcg - Advair Diskus 100/50 mcg

2. Secondary Outcome: Change From Baseline at 12 Hours Post-Dose in Forced Expiratory Volume in One Second (FEV1) By Treatment
Description: The secondary efficacy variable was the change from period-specific baseline in FEV1 at 12 hours, calculated as FEV1 measured at 12 hours postdose after subtracting period-specific baseline FEV1 at each treatment period.
  The period-specific baseline FEV1 was measured at predose within 5 minutes of AM dose administration at each treatment visit. If that value was missing, then FEV1 measured at 30 minutes predose was used as the period-specific baseline.
Time Frame: Pre-dose: 30 minutes prior, within 5 minutes of dose. Post-dose: 12 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg
Number analyzed (Participants) | 67 | 67 | 68 | 67 | 68 | 66
mL | 11.53 (29.058) | 128.49 (29.109) | 170.51 (28.990) | 209.85 (29.127) | 238.30 (28.988) | 170.54 (29.230)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/50 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/50 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 226.77, 95% CI 2-sided [172.4 to 281.1] — FS MDPI 100/50 mcg - Fp MDPI 100 mcg
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/25 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/25 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 198.32, 95% CI 2-sided [143.7 to 252.9] — FS MDPI 100/25 mcg - Fp MDPI 100 mcg
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/12.5mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/12.5 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 158.99, 95% CI 2-sided [104.7 to 213.3] — FS MDPI 100/12.5 mcg - Fp MDPI 100 mcg
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs FS MDPI 100/6.25 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/6.25 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 116.96, 95% CI 2-sided [62.4 to 171.6] — FS MDPI 100/6.25 mcg - Fp MDPI 100 mcg
Statistical Analysis 5: Comparison: Fp MDPI 100 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each Advair Diskus 100/50 mcg dose group and Fp MDPI 100 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 159.01, 95% CI 2-sided [104.3 to 213.7] — Advair Diskus 100/50 mcg - Fp MDPI 100 mcg
Statistical Analysis 6: Comparison: FS MDPI 100/50 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/50 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.0150, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 67.76, 95% CI 2-sided [13.3 to 122.2] — FS MDPI 100/50 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 7: Comparison: FS MDPI 100/25 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/25 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.1578, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 39.31, 95% CI 2-sided [-15.3 to 94.0] — FS MDPI 100/25 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 8: Comparison: FS MDPI 100/12.5mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/12.5 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.9993, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = -0.02, 95% CI 2-sided [-54.4 to 54.4] — FS MDPI 100/12.5 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 9: Comparison: FS MDPI 100/6.25 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each FS MDPI 100/6.25 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p = 0.1311, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = -42.05, 95% CI 2-sided [-96.7 to 12.6] — FS MDPI 100/6.25 mcg - Advair Diskus 100/50 mcg
Statistical Analysis 10: Comparison: Fp MDPI 100 mcg vs Advair Diskus 100/50 mcg; The estimated treatment difference from the ANCOVA model between each Fp MDPI 100 mcg dose group and Advair Diskus 100/50 mcg group is presented together with the two-sided 95% CI for the difference and the p-value; Test type: Superiority; p < 0.0001, ANCOVA — significance of 0.05 or alpha of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = -159.01, 95% CI 2-sided [-213.7 to -104.3] — Fp MDPI 100 mcg - Advair Diskus 100/50 mcg

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC0-t) of Salmeterol
Description: Blood samples for measurement of plasma SAL concentrations were obtained during each treatment visit (subjects 18 years of age and older only) and pharmacokinetic parameters were derived. The primary pharmacokinetic parameters were AUC0-t and Cmax for Salmeterol.
Time Frame: Predose (0), and at 5, 10, 15 and 30 minutes, 1, 1.5, 2, 3, 4, 8, and 12 hours postdose
Population: Pharmacokinetic Analysis set. PK parameters for Salmeterol were not run for Fp MDPI experience.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg
Number analyzed (Participants) | 0 | 62 | 65 | 61 | 61 | 62
pg*hr/mL |  | 32.8 (20.98) | 69.9 (35.36) | 133.5 (63.13) | 309.3 (143.43) | 173.5 (106.59)
Statistical Analysis 1: Comparison: FS MDPI 100/50 mcg vs Advair Diskus 100/50 mcg; The analysis is based on ANOVA model of the log transformed data, with fixed effects of sequence, period and treatment, and a random effect for subject within sequence. n=58; Test type: Superiority; geometric mean ratio = 1.929, 90% CI 2-sided [1.690 to 2.202]
Statistical Analysis 2: Comparison: FS MDPI 100/25 mcg vs Advair Diskus 100/50 mcg; The analysis is based on ANOVA model of the log transformed data, with fixed effects of sequence, period and treatment, and a random effect for subject within sequence. n=59; Test type: Superiority; geometric mean ratio = 0.800, 90% CI 2-sided [0.702 to 0.911]
Statistical Analysis 3: Comparison: FS MDPI 100/12.5mcg vs Advair Diskus 100/50 mcg; The analysis is based on ANOVA model of the log transformed data, with fixed effects of sequence, period and treatment, and a random effect for subject within sequence. n=61; Test type: Superiority; geometric mean ratio = 0.427, 90% CI 2-sided [0.376 to 0.485]
Statistical Analysis 4: Comparison: FS MDPI 100/6.25 mcg vs Advair Diskus 100/50 mcg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; LSM difference = 0.172, 90% CI 2-sided [0.151 to 0.196]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Salmeterol
Description: as for outcome 3
Time Frame: Predose (0), and at 5, 10, 15 and 30 minutes, 1, 1.5, 2, 3, 4, 8, and 12 hours postdose
Population: Pharmacokinetic Analysis set. PK parameters for Salmeterol were not run for Fp MDPI experience.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg
Number analyzed (Participants) | 0 | 62 | 65 | 61 | 61 | 62
pg/mL |  | 16.0 (8.86) | 35.8 (20.25) | 67.5 (34.71) | 154.5 (80.28) | 42.3 (19.28)
Statistical Analysis 1: Comparison: FS MDPI 100/50 mcg vs Advair Diskus 100/50 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; geometric mean ratio = 3.622, 90% CI 2-sided [3.149 to 4.168]
Statistical Analysis 2: Comparison: FS MDPI 100/25 mcg vs Advair Diskus 100/50 mcg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; geometric mean ratio = 1.534, 90% CI 2-sided [1.335 to 1.763]
Statistical Analysis 3: Comparison: FS MDPI 100/12.5mcg vs Advair Diskus 100/50 mcg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; geometric mean ratio = 0.795, 90% CI 2-sided [0.694 to 0.911]
Statistical Analysis 4: Comparison: FS MDPI 100/6.25 mcg vs Advair Diskus 100/50 mcg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; geometric mean ratio = 0.339, 90% CI 2-sided [0.295 to 0.390]

5. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Salmeterol
Description: Blood samples for measurement of plasma SAL concentrations were obtained during each treatment visit (subjects 18 years of age and older only) and pharmacokinetic parameters were derived.
Time Frame: Predose (0), and at 5, 10, 15 and 30 minutes, 1, 1.5, 2, 3, 4, 8, and 12 hours postdose
Population: Pharmacokinetic Analysis set. PK parameters for Salmeterol were not run for Fp MDPI experience.
Measure: Median (Full Range); unit: hours
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg
Number analyzed (Participants) | 0 | 62 | 65 | 61 | 61 | 62
hours |  | 0.1 [0.1 to 12.1] | 0.1 [0.1 to 2.0] | 0.1 [0.1 to 2.0] | 0.1 [0.1 to 1.5] | 0.5 [0.1 to 2.0]

6. Secondary Outcome: Patients With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: TEAEs were recorded during each double-blind treatment. In addition, at the end of each treatment, patients continued to use 2 inhalations of Fp MDPI 50 mcg (100 mcg total dose) twice daily, so adverse events during this treatment were assigned to Fp MDPI 50 mcg.
  An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical in
Time Frame: Day 1 up to Day 35
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Fp MDPI 50 mcg X 2 BID: Patients used 2 inhalations of Fp MDPI 50 mcg (100 mcg total dose) twice daily during the 'washout' between treatment periods, so adverse events during this treatment were assigned to Fp MDPI 50 mcg.
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg | Fp MDPI 50 mcg X 2 BID
Number analyzed (Participants) | 67 | 68 | 69 | 67 | 68 | 66 | 72
Participants
  Any adverse event | 2 | 2 | 3 | 1 | 1 | 3 | 17
  Severe adverse event | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Treatment-related adverse event | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Withdrawn from treatment due to AE | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 35
Arm/Group | Fp MDPI 100 mcg | FS MDPI 100/6.25 mcg | FS MDPI 100/12.5mcg | FS MDPI 100/25 mcg | FS MDPI 100/50 mcg | Advair Diskus 100/50 mcg | Fp MDPI 50 mcg X 2 BID
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68 | 0/69 | 0/67 | 0/68 | 0/66 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68 | 0/69 | 0/67 | 0/68 | 0/66 | 0/72
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68 | 0/69 | 0/67 | 0/68 | 0/66 | 4/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fp MDPI 100 mcg (N=67) | FS MDPI 100/6.25 mcg (N=68) | FS MDPI 100/12.5mcg (N=69) | FS MDPI 100/25 mcg (N=67) | FS MDPI 100/50 mcg (N=68) | Advair Diskus 100/50 mcg (N=66) | Fp MDPI 50 mcg X 2 BID (N=72)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.